CLINICAL TRIAL: NCT05881512
Title: Early Feasibility Study of Transcutaneous Upper Airway Stimulation in Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somnial Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SOMN-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea; OSA
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- TUAS (Experimental): Transcutaneous upper airway stimulation
  Interventions: Device: Transcutaneous Upper Airway Stimulation Device

INTERVENTIONS:
Device: Transcutaneous Upper Airway Stimulation Device — Multiple frequency stimulation of the hypoglossal nerve
  Other Names: TUAS

SUMMARY:
Early feasibility study to estimate the functionality of a novel intervention based on non-invasive transcutaneous electrical stimulation of the hypoglossal nerve to reduce the Apnea Hypopnea Index (AHI).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years or older
* In good general health, as evidenced by medical history and diagnosed with moderate or severe OSA
* In-lab PSG, within the last 6 months, with an AHI of 15-50/hour. In addition, <25% of the respiratory events on the diagnostic PSG can be attributed to central apneas
* BMI less than or equal to 32

Exclusion Criteria:

* No or mild OSA (AHI <15/h) or very severe OSA (AHI >50/hour), exclusively postural sleep apnea, or isolated Rapid-Eye-Movement (REM) sleep associated OSA.
* Patients who are cachectic (BMI <18.5 kg/m2) or obese (BMI >32 kg/m2).
* Patients should not have enlarged tonsils (size 3-4) and/or adenoids, nasal polyps, neuromuscular disease, hypoglossal nerve palsy, abnormal pulmonary function tests, severe pulmonary hypertension, valvular heart disease, heart failure (New York Heart Association, NYHA III-IV), recent myocardial infarction, significant cardiac arrhythmias, atrial fibrillation, stroke, opioid usage, uncontrolled hypertension, known allergic reaction to adhesives or latex, active psychiatric disease, co-existing non-respiratory sleep disorder, pregnancy or significant metal implants or cardiac/other pacemakers.
* Patients with facial hair that affects the correct placement of the electrodes, if they are unwilling to shave.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | Overnight (day 1)
  Episodes of apnea and/or hypopnea scored during the course of sleep study

SECONDARY OUTCOMES:
Arterial Oxygen Saturation (SaO2) | Overnight (day 1)
  SaO2 levels during the course of sleep study compared to baseline

OTHER OUTCOMES:
Sleep Quality | Overnight (day 1)
  Subjective Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lee Shangold, MD, Principal Investigator — ENT & Allergy Associates, LLP
Locations (1):
- United Diagnostics, Commack, New York, United States